CLINICAL TRIAL: NCT05080725
Title: Measuring Pharyngeal Muscle Improvements Following Behavioral Swallowing Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-00860
Record Dates: First submitted 2021-09-09; First posted 2021-10-18 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Generalized sarcopenia group (Experimental): Older adults will be recruited from local community centers, physician offices, and retirement communities via flyers. Participants will complete 16 sessions of standard of care swallowing exercises 2 times per week for 8 weeks. All sessions will be conducted via Webex. During each session, a series of standard of care swallow exercises will be performed following a demonstration from a trained speech-language pathologist.
  Interventions: Other: TelePEPP intervention

INTERVENTIONS:
Other: TelePEPP intervention — TelePEPP sessions will be conducted twice per week by a Speech Language Pathologist and/or graduate student clinician, on the study team. This clinician will deliver the intervention from the NYU Voice Center using the web conferencing software Webex (institutional license) on a Dell desktop computer with a 3.1 GHz intel core processor and high definition camera. Each exercise set will include 40 repetitions (10 reps of effortful swallows, tongue hold swallows, effortful pitch glides and maximal posterior tongue presses). All exercises are widely-adopted by clinicians as standard of care exercises. The number of sets will be gradually increased as tolerance builds [2 sets in week 1, 3 sets in week 2, 4 sets in weeks 3+].

SUMMARY:
The purpose of this study is to learn more about how exercise and protein supply affect swallow muscles. Twenty healthy older adults will be recruited from local community centers, physician offices, and retirement communities via flyers. Participants will complete 16 sessions of standard of care swallowing exercises 2 times per week for 8 weeks. All sessions will be conducted via Zoom. During each session, a series of swallow exercises will be performed following a demonstration from a trained speech-language pathologist. Participants will be referred to NYU Langone Health or White Plains Hospital, for a videofluoroscopic swallowing study, acoustic pharyngometry and measures of hand grip strength before and after the treatment protocol. Patients will be able to select their preferred site for swallow study completion. Results will inform the relationship between swallow exercises and pharyngeal muscles. All devices and exercises are established as safe and effective and are FDA approved.

DETAILED DESCRIPTION:
The natural next step in this program of research is to investigate interventions for reversing pharyngeal sarcopenia with the ultimate goal of developing novel therapeutic strategies to address this pervasive clinical issue. The exercise science literature suggests that sarcopenia in the limb muscles can be reversed through a combination of rigorous exercise and adequate levels of dietary protein. The innovative multi-disciplinary protocol, PEPP (Pharyngeal Exercises Plus Protein), combines pharyngeal swallowing exercises selected for their known activation of the pharyngeal muscles with daily supplemental protein drinks. The research lab had documented successful improvements to swallowing physiology and pharyngeal sarcopenia in a pilot series of 5 older women using PEPP. However the research was abruptly halted due to both ethical and feasibility challenges posed by the COVID-19 pandemic. In response to these challenges, this study is seeking to establish the feasibility and effectiveness when the PEPP intervention is delivered using telehealth (telePEPP).

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* SARC-F score of ≥4
* Functional hearing and vision status
* Access to reliable internet connection
* Availability of caregiver/family support and/or comfort with independent technology usage

Exclusion Criteria:

* Known structural or neurological causes of dysphagia
* Not suitable to consume high levels of protein supplementation (i.e. moderate to severe kidney dysfunction)

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Measurement of pharyngeal constriction before intervention | Session 0 (Day 0 pre-intervention visit)
  2D lateral videofluoroscopic images will be used to measure pharyngeal constriction pre and post intervention
Measurement of pharyngeal constriction after intervention | Session 17 (9 week post-intervention visit)
  2D lateral videofluoroscopic images will be used to measure pharyngeal constriction pre and post intervention
Measurement of pharyngeal shortening before intervention | Session 0 (Day 0 pre-intervention visit)
  2D lateral videofluoroscopic images will be used to measure pharyngeal shortening pre and post intervention
Measurement of pharyngeal shortening after intervention | Session 17 (9 week post-intervention visit)
  2D lateral videofluoroscopic images will be used to measure pharyngeal shortening pre and post intervention

SECONDARY OUTCOMES:
Measurement of pharyngeal wall thickness before intervention | Session 0 (Day 0 pre-intervention visit)
  2D lateral videofluoroscopic images will be used to measure wall thickness pre and post intervention
Measurement of pharyngeal wall thickness after intervention | Session 17 (9 week post-intervention visit)
  2D lateral videofluoroscopic images will be used to measure wall thickness pre and post intervention
Measurement of pharyngeal volume before intervention | Session 0 (Day 0 pre-intervention visit)
  Acoustic Pharyngometry will be used to measure pharyngeal volume pre and post intervention.
Measurement of pharyngeal volume after intervention | Session 17 (9 week post-intervention visit)
  Acoustic Pharyngometry will be used to measure pharyngeal volume pre and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja M Molfenter, PhD, CCC-SLP, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This study is to collect a series of pilot data to support an NIH grant submission to test the intervention during a randomized control trial. If the application is successful, the IPD of the NIH funded RCT will be made sharable.